CLINICAL TRIAL: NCT05265871
Title: ATP Level in Induced Sputum and Cough Sensitivity to ATP in Subjects With Refractory/Unexplained Chronic Cough
Brief Title: ATP Level and Cough Sensitivity to ATP in Subjects With Refractory/Unexplained Chronic Cough
Status: Completed | Type: Observational
Sponsor: Kefang Lai (Other)
Responsible Party: Sponsor-Investigator, Kefang Lai, Director of Clinical Research Department, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: RCC-ATP
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Refractory/Unexplained Chronic Cough
Keywords: refractory/unexplained chronic cough; cough sensitivity; adenosine triphosphate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — sputum supernate (without DNA)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- refractory/unexplained chronic cough: Induced sputum test and cough challenge(ATP and capsaicin) were performed.
- Healthy control: Induced sputum test and cough challenge(ATP and capsaicin ) were performed.

SUMMARY:
This is a cross-sectional study to investigate ATP level in induced sputum and cough sensitivity to ATP in subjects with refractory/unexplained chronic cough. 60 patients with refractory/unexplained chronic cough and 30 matched healthy controls were recruited. Demographic data, clinical characteristic, cough sacles and medical history records were collected. Cough chanllage(ATP and capsaicin) and ATP measurement in sputum were conducted.The difference of sputum ATP level between patients and control and the correlation between sputum ATP level and cough sensitivity to ATP were analyzed.

ELIGIBILITY:
Inclusion criteria for patients:

1. ≥18 years old
2. cough as sole symptom lasting ≥6 months
3. cough visual analogue score ≥30mm
4. diagnosed as RCC/UCC according to guidelines

Exclusion criteria for patients:

1. smoking currently or in the past 6 months, or a smoking history of >20 pack-year
2. a forced expiratory volume in 1 second/forced vital capacity ratio <70%;
3. use of inhaled/oral corticosteroid, bronchodilators, anti-allergic medicine, antitussive medicine or anti-reflux treatment in the past 1 week;
4. a history of acute respiratory infection in the past 4 weeks;
5. a history of severe disease (cancer, acute coronary syndrome and so on).

Healthy control aged ≥18 years old are included. Exclusion criteria are as follow:

1. smoking currently or in the past 6 months, or a smoking history of >20 pack-year
2. a forced expiratory volume in 1 second/forced vital capacity ratio <70%
3. a history of acute respiratory infection in the past 4 weeks
4. posstive findings of chest radiography
5. a history of chronic respiratory disease and allergic disease
6. any signs of cough hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic cough visiting cough clinics at the First Affiliated Hospital of Guangzhou Medical University would all be screened by the investigator. To be specific, RCC/UCC refers to a chronic cough: 1) without identifiable causes after throughout investigation; 2) persistent after empirical treatment to known causes; 3) persistent after treatment for positive conditions known to be associated with chronic cough. Age and gender matched healthy controls would be recruited.
  The subject who meets the criteria and provides written informed consent is considered as eligible and enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kefang Lai, MD, PhD, Study Chair — Guangzhou Institute of Respiratory Health, State Key Laboratory of Respiratory Disease, National Clinical Research Center for Respiratory Disease, National Center for Respiratory Medicine, The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Institute of Respiratory Health, State Key Laboratory of Respiratory Disease, National Clinical Research Center for Respiratory Disease, National Center for Respiratory Medicine, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Refractory/Unexplained Chronic Cough: Patients with RCC/UCC were recruited in the Cough Clinic at the First Affiliated Hospital of Guangzhou Medical University from May 2022 to January 2024. To be specific, RCC/UCC refers to a chronic cough: 1) without identifiable causes after throughout investigation; 2) persistent after empirical treatment to known causes; 3) persistent after treatment for positive conditions known to be associated with chronic cough.
  Inclusion criteria for patients:
  1. ≥18 years old
  2. cough as sole symptom lasting ≥6 months
  3. cough visual analogue score ≥30mm
  4. diagnosed as RCC/UCC according to guidelines
  Exclusion criteria for patients:
  1. smoking currently or in the past 6 months, or a smoking history of >20 pack-year
  2. a forced expiratory volume in 1 second/forced vital capacity ratio <70%;
  3. use of inhaled/oral corticosteroid, bronchodilators, anti-allergic medicine, antitussive medicine or anti-reflux treatment in the past 1 week;
  4. a history of acute respiratory infection in the past 4 weeks;
  5. a history of severe disease (cancer, acute coronary syndrome and so on).
- Healthy Controls: Healthy control (≥18 years old) are included, who are age and gender marched with patients. Exclusion criteria are as follow:
  1. smoking currently or in the past 6 months, or a smoking history of >20 pack-year
  2. a forced expiratory volume in 1 second/forced vital capacity ratio <70%
  3. a history of acute respiratory infection in the past 4 weeks
  4. posstive findings of chest radiography
  5. a history of chronic respiratory disease and allergic disease
  6. any signs of cough hypersensitivity
Period: Overall Study
Arm/Group | Patients With Refractory/Unexplained Chronic Cough | Healthy Controls
Started | 101 | 30
Completed | 101 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Refractory/Unexplained Chronic Cough | Healthy Controls | Total
Number analyzed (Participants) | 101 | 30 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.1) | 42.6 (10.8) | 40.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 14 | 68
  Male | 47 | 16 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 101 | 30 | 131
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: ATP Level in Sputum Supernatant
Description: ATP level in induced sputum in patients with refractory/unexplained chronic cough and healthy control
Time Frame: ATP concentrations were measured in all specimens on the day of the last participant's enrollment.
Measure: Mean (Inter-Quartile Range); unit: pM
Groups:
- Patients With Refractory/Unexplained Chronic Cough: Induced sputum test and cough challenge(ATP and capsaicin) were performed.
Arm/Group | Patients With Refractory/Unexplained Chronic Cough | Healthy Control
Number analyzed (Participants) | 96 | 25
pM | 2313.4 [1312.3 to 4633.8] | 1804.6 [1237.3 to 5276.2]

2. Secondary Outcome: ATP Cough Sensitivity
Description: Cough sensitivity for ATP in patients with refractory/unexplained chronic cough and healthy control. Lowest concentration of ATP that provoked at least 5 coughs (C5) is used to indicate cough sensitivity.
Time Frame: Each subject underwent ATP cough challenge on the day of enrollment.
Measure: Mean (Inter-Quartile Range); unit: mM
Arm/Group | Patients With Refractory/Unexplained Chronic Cough | Healthy Control
Number analyzed (Participants) | 101 | 30
mM | 3.16 [0.316 to 31.6] | 316 [31.6 to 316]

ADVERSE EVENTS:
Time Frame: This study mainly involves induced sputum test and cough challenge without any interventional design. Induced sputum test and cough challenge are received as safe and widely used in clinics or researches. Therefore, observation of adverse event has not been designed.
Description: All-Cause mortality, serious, and other [Not Including Serious] adverse events were not monitored, so total number of participants at risk for adverse events is zero.
Arm/Group | Patients With Refractory/Unexplained Chronic Cough | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT05265871/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT05265871/SAP_001.pdf